CLINICAL TRIAL: NCT02949778
Title: Quadratus Lumborum Block for Perioperative Analgesia in Patients Treated With Abdominoplasty: A Randomised Controlled Trial
Brief Title: Quadratus Lumborum Block for Abdominoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BS-AIO-2015-QL-block
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Pain, Postoperative; Abdominoplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine 3.75mg/mL (Active Comparator): QL-block using 20 mL ropivacaine 3.75mg/mL
  Interventions: Procedure: QL-block; Drug: Ropivacaine
- Sodium chloride 9 mg/mL (Placebo Comparator): QL-block using 20 mL sterile sodium chloride 9 mg/mL
  Interventions: Procedure: QL-block; Drug: Sodium Chloride

INTERVENTIONS:
Procedure: QL-block — Bilateral quadratus lumborum block using either ropivacaine 3.75mg/ml or sodium chloride 0.9% is the intervention studied
  Other Names: Quadratus lumborum block
Drug: Ropivacaine — Ropivacaine 3.75mg/ml administered in QL-block as active treatment
  Other Names: Naropin
  Arms: Ropivacaine 3.75mg/mL
Drug: Sodium Chloride — Sodium chloride 9mg/mL administered in QL-Block as placebo
  Arms: Sodium chloride 9 mg/mL

SUMMARY:
Double blinded, randomized, controlled, phase IV intervention trial. Both groups will receive a quadratus lumborum Block (QL), using ropivacaine 3.75 mg/mL in the intervention group, and sterile sodium chloride in the control group. The aim of study is to investigate the effect of a QL Block on the perioperative pain during postbariatric abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Classification Status (ASA) I-II
* Age 18 to 64
* Weight above or equal to 60 kg
* Scheduled for post-bariatric surgery with standard full abdominoplasty performed by Dr Frøyen
* Patient is expected able to cooperate during the treatment and follow up.
* Signed informed consent obtained and documented according to the International Conference on Harmonization (ICH) good clinical practice (GCP), and national/local regulations.

Exclusion Criteria:

* A history of anaphylactic shock
* Cardiovascular disease other than hypertension and/or hyperlipidemia
* Known allergy to ropivacaine or morphine
* A history of chronic pain
* Psychiatric comorbidity
* Scheduled opioid pain medication or neuroleptic drugs
* Coagulation disorders or treatment with platelet inhibitors
* Pregnancy or breastfeeding
* Treatment with class III antiarrhythmics, sertindole, ziprasidone, amisulpride, ceritinib, hydroxyzine, fluvoxamine
* Any medical contraindication to the study intervention by the attending anaesthetist or surgeon (to be specified in screening form).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  total opioid consumption the first 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Thor Wilhelm Bjelland, MD, PhD, Principal Investigator — Vestre Viken HT, Baerum Hospital
Locations (1):
- Vestre Viken HT, Baerum Hospital, Sandvika, Norway

IPD SHARING:
Plan to Share IPD: No
Requires approval by ethics committee and second consent form.